CLINICAL TRIAL: NCT03041415
Title: Citizen Science to Promote Sustained Physical Activity in Low-Income Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Abby C King, Professor of Health Research & Policy and Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA211048 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-02-02 (Estimated); Results first posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-04

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: group-randomized design to either a person-level physical activity intervention alone, or the person-level physical activity intervention plus a citizen science intervention aimed at making the local neighborhood more activity-supportive.
Who Masked: Outcomes Assessor
Masking Description: Assessors will not be told the intervention assigned of the participating housing sites
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALED Alone Physical Activity Program (Active Comparator): * The Active Living Every Day (ALED) comprehensive 12-week PA training and support program is appropriate for delivery by trained instructors from diverse backgrounds.
  * Participants are taught self-regulatory skills aimed at increasing and sustaining regular physical activities such as walking.
  Interventions: Behavioral: ALED Alone Physical Activity Program
- ALED + Our Voice PA Program (Experimental): * The ALED physical activity program is combined with the Our Voice citizen science engagement program, which teaches participants how to assess the barriers and enablers of neighborhood physical activity using a simple mobile app.
  * Residents then share their data and build consensus around major barriers and potential solutions, which they share with local decision makers.
  Interventions: Behavioral: ALED + Our Voice PA Program

INTERVENTIONS:
Behavioral: ALED Alone Physical Activity Program — • 12-week class focused on teaching self-regulatory skills to increase regular PA
  Arms: ALED Alone Physical Activity Program
Behavioral: ALED + Our Voice PA Program — * 12-week class focused on teaching self-regulatory skills to increase regular PA
  * Neighborhood assessment, consensus-building, & advocacy program in which participants are taught skills to promote neighborhood-level changes in support of regular Physical activity
  Arms: ALED + Our Voice PA Program

SUMMARY:
While low-income midlife and older adults are disproportionately affected by chronic diseases that can be alleviated by regular physical activity, few physical activity programs have been developed specifically with their needs in mind. Those programs that are available typically do not address the recognized local environmental factors that can impact physical activity. This research aims to evaluate the added effects on two-year physical activity levels of a novel citizen science neighborhood engagement program (called Our Voice) when combined with an evidence-based, individually-focused physical activity program (Active Living Every Day), relative to the individually-focused program alone. The programs will be delivered in affordable housing settings, and represent a potentially scalable means for promoting physical activity across broader income groups in the US.

DETAILED DESCRIPTION:
The major objective of this project is to enhance the potential scalability and sustainability of person-level physical activity (PA) interventions by leveraging the capacity of residents themselves as local data gatherers and solution generators for neighborhood environmental change. The primary aim of the group-randomized trial is to systematically compare the sustained (two-year) multi-level impacts of a lay advisor-delivered, person-level PA intervention that has demonstrated efficacy and translatability (Active Living Every Day) [ALED Alone arm], versus the ALED program in combination with a novel neighborhood-level intervention, called Our Voice [ALED+Our Voice arm]. The Our Voice program teaches residents to use a simple mobile application to individually and collectively identify neighborhood barriers to daily PA. They then convey this information to local stakeholders and decision-makers in ways that can facilitate potentially sustainable neighborhood-level improvements in support of regular PA. Up to sixteen affordable housing sites serving low-income, ethnically diverse midlife and older adults will be randomized to one of the two interventions.

ELIGIBILITY:
Inclusion Criteria:

* Lives in or around a designated housing site;
* Is insufficiently physically active based on National guidelines;
* Can engage in moderate forms of PA such as walking;
* No plans to move from the area over the 2-year period;
* Willing to engage in study assessments.

Exclusion Criteria:

* Only one eligible member of a household will be enrolled;
* Medical conditions which contraindicate participation in regular, unsupervised moderate-intensity physical activity.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Commensurate with current requirements, once the study data have undergone final data cleaning, analysis, and planned publication, the investigators will make the final data collected as part of the proposed research available in electronic form to researchers who request them. The investigators will request that researchers submit a data request in writing to the project principal investigator so that the requested data can be made available while protecting the confidentiality of study participants. By setting up a centralized data request process, the investigators will be able to provide requestors with information that will help to inform external research groups about duplicate data analysis activities on the part of other research groups related to the data set in question.

REFERENCES:
- [Background] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760
- [Derived] King AC, Campero MI, Garcia D, Blanco-Velazquez I, Banchoff A, Fierros F, Escobar M, Cortes AL, Sheats JL, Hua J, Chazaro A, Done M, Espinosa PR, Vuong D, Ahn DK. Testing the effectiveness of community-engaged citizen science to promote physical activity, foster healthier neighborhood environments, and advance health equity in vulnerable communities: The Steps for Change randomized controlled trial design and methods. Contemp Clin Trials. 2021 Sep;108:106526. doi: 10.1016/j.cct.2021.106526. Epub 2021 Aug 8. PMID 34371162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in groups/clusters (affordable housing sites) to receive the assigned interventions.
Units Other Than Participants: Affordable housing sites
Groups:
- ALED Alone Physical Activity (PA) Program: * The Active Living Every Day (ALED) comprehensive 12-week PA training and support program is appropriate for delivery by trained instructors from diverse backgrounds.
  * Participants are taught self-regulatory skills aimed at increasing and sustaining regular physical activities such as walking.
  ALED Alone Physical Activity Program: • 12-week class focused on teaching self-regulatory skills to increase regular PA
- ALED + Our Voice PA Program: * The ALED physical activity program is combined with the Our Voice citizen science engagement program, which teaches participants how to assess the barriers and enablers of neighborhood physical activity using a simple mobile app.
  * Residents then share their data and build consensus around major barriers and potential solutions, which they share with local decision makers.
  ALED + Our Voice PA Program: • 12-week class focused on teaching self-regulatory skills to increase regular PA
  • Neighborhood assessment, consensus-building, & advocacy program in which participants are taught skills to promote neighborhood-level changes in support of regular Physical activity
Period: Overall Study
Arm/Group | ALED Alone Physical Activity (PA) Program | ALED + Our Voice PA Program
Started | 140; 5 Affordable housing sites | 160; 5 Affordable housing sites
Completed | 123; 5 Affordable housing sites | 145; 5 Affordable housing sites
Not Completed | 17; 0 Affordable housing sites | 15; 0 Affordable housing sites

BASELINE CHARACTERISTICS:
Groups:
- ALED Alone Physical Activity Program: * The Active Living Every Day (ALED) comprehensive 12-week PA training and support program is appropriate for delivery by trained instructors from diverse backgrounds.
  * Participants are taught self-regulatory skills aimed at increasing and sustaining regular physical activities such as walking.
  ALED Alone Physical Activity Program: • 12-week class focused on teaching self-regulatory skills to increase regular PA
- Total: Total of all reporting groups
Arm/Group | ALED Alone Physical Activity Program | ALED + Our Voice PA Program | Total
Number analyzed (Participants) | 140 | 160 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 92
  >=65 years | 92 | 116 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.04 (10.91) | 69.93 (9.74) | 69.52 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 119 | 221
  Male | 38 | 41 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 36 | 55
  Not Hispanic or Latino | 121 | 124 | 245
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 28 | 27 | 55
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 87 | 88 | 175
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 36 | 55
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 140 | 160 | 300

OUTCOME MEASURES:

1. Primary Outcome: Weekly Walking Minutes
Description: Self-report using the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire. CHAMPS is a self-report physical activity questionnaire that assesses weekly frequency and duration of various activities typically undertaken by midlife and older adults over the prior 4-week period. Self-reported walking for errands is one physical activity item assessed. The measure has been shown to have good test-retest reliability (stability) and construct and concurrent validity, and has been shown to be sensitive to change in a variety of adult populations. It has seven frequency categories (from less than 1 hour a week to 9 or more hours per week). The minimum value is 0 and the maximal value is variable.
Time Frame: 12 months
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | ALED Alone Physical Activity Program | ALED + Our Voice PA Program
Number analyzed (Participants) | 123 | 145
minutes/week | 189.5 (227.7) | 206.7 (198.7)

2. Secondary Outcome: Total Physical Activity
Description: as for outcome 1
Time Frame: 12 months
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | ALED Alone Physical Activity Program | ALED + Our Voice PA Program
Number analyzed (Participants) | 123 | 145
minutes/week | 596.2 (443.9) | 562.0 (389.2)

3. Secondary Outcome: Moderate-to-Vigorous Physical Activity
Description: Self-report using the Community Healthy Activities Model Program for Seniors (CHAMPS) Physical Activity Questionnaire, supported via accelerometer (Actigraph). CHAMPS is A self-report physical activity questionnaire that assesses weekly frequency and duration of various activities typically undertaken by midlife and older adults over the prior 4-week period. Self-reported walking for errands is one physical activity item assessed. The measure has been shown to have good test-retest reliability (stability) and construct and concurrent validity, and has been shown to be sensitive to change in a variety of adult populations. It has seven frequency categories (from less than 1 hour a week to 9 or more hours per week). The minimum value is 0 and the maximal value is variable.
Time Frame: 12 months
Population: Participants who completed the protocol are included in the analysis
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | ALED Alone Physical Activity Program | ALED + Our Voice PA Program
Number analyzed (Participants) | 123 | 145
minutes/week | 117.4 (232.6) | 108.8 (139.4)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | ALED Alone Physical Activity Program | ALED + Our Voice PA Program
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/160
Other Adverse Events (participants affected / at risk) | 0/140 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT03041415/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT03041415/SAP_001.pdf
  • Informed Consent Form (2019-08-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT03041415/ICF_002.pdf